CLINICAL TRIAL: NCT03135873
Title: Mastiha Treatment for Obese With NAFLD Diagnosis
Acronym: MAST4HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: University of Novi Sad (Other); National Research Council, Institute of Clinical Physiology, Italy (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Assistant Professor in Foods and Human Nutrition, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAST4HEALTH (691042)
Record Dates: First submitted 2017-03-09; First posted 2017-05-01 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — mastiha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mastiha (Active Comparator): This arm of patients will receive natural Mastiha supplements at a daily dosage of 2.1 g for a 6 month period.
  Interventions: Dietary Supplement: Mastiha
- Placebo (Placebo Comparator): This arm of patients will receive placebo for a 6 month period.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mastiha — Mastiha is a natural product of Greece and has a license of manufactures Foods for Particular Nutritional Uses and of National Organization of Medicines (EOF).
  Arms: Mastiha
Dietary Supplement: Placebo — Placebo is designed to have identical characteristics with verum.
  Arms: Placebo

SUMMARY:
NAFLD/NASH is one of the most common complications of obesity and diabetes mellitus in Western populations affecting approximately 50% of diabetics and 76% of obese patients. Due to the lack of specialized treatment, many new efforts focus on exploring alternative, non-pharmacologic means for managing the disease, including bioactive substances in fruits, vegetables and plants or their products. Mastiha, a natural product of Greece, consists of a great variety of bioactive phytochemical compounds and demonstrates antioxidant, antiinflammatory, antimicrobial and lipid lowering properties. Taking into account the contribution of oxidative stress and inflammation to NAFLD/NASH pathogenesis, the hypothesis that Mastiha could improve disease aspects is investigated. Thus, design of a multicenter (4 centers across Europe), randomized, double-blind, placebo controlled (parallel arm) clinical trial to assess the effect of Mastiha on clinical course of NAFLD/NASH patients has been conducted. The effectiveness of the proposed intervention will be evaluated via clinical and laboratory markers. MAST4HEALTH aims also at exploring gene-diet interactions and at correlating genetic and epigenetic markers with metabolomic and intestinal microbiota profiles pre- and post- intervention. To this end, patients with confirmed NAFLD/NASH will be allocated to either verum or placebo group. Duration of the intervention will be 6 months and the dosage applied will be 2.1 g daily. NAFLD/NASH diagnosis will be confirmed by MS scanning and the sensitive LiverMultiScan technique. Anthropometric, demographic data, body composition, dietary habits, physical activity, family history and smoking status will be assessed pre- and post- intervention. Biochemical profile, oxidative stress and inflammation, as well as epigenetic and metabolomic profiles will be assessed in blood samples, while the metagenome profile will be examined in stools. Both groups will receive counselling to allow for body weight regulation up to 5%. Compliance will be assessed monthly and side effects will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed NAFLD/NASH
* 18 years < Age < 67 years
* BMI > 30 kg/ m2

Exclusion Criteria:

* Hepatotoxic Medication, Concomitant Liver Disease
* Decompensated Diabetes Mellitus
* Dysthyroidism, hypopituitarism, Cushing syndrome / disease
* Alcohol abuse or drug addiction
* Clinically or biochemically recognized systemic diseases
* Pregnancy test, lactation
* Vegan or lacto- and ovo-lacto- vegetarianism
* Psychiatric or mental disorder
* Recent loss in body weight or current diet
* Any use of antioxidant-phytochemical rich supplement, anti-, pre- or pro-biotics within 3 months pre-intervention
* Changes in drug treatment for e.g. hypertension, diabetes mellitus, 3 months prior or during the 6month intervention
* Antibiotic treatment during and 2 months prior to screening

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
LIF score | 6 months
  Improvement in liver histopathology reflected in reduction of the sensitive LIF score

SECONDARY OUTCOMES:
NAFLD/NASH-related laboratory markers | 6 months
  Liver enzymes improvement, inflammation and oxidative stress markers improvement (e.g. IL-6, IL-10, TNF-α, GSH, Gpx), lipid profile improvement, insulin sensitivity improvement pre- and post- intervention in each intervention arm.
Anthropometric characteristics | 6 months
  BMI pre- and post- intervention in each intervention arm.
Genetic profile | 6 months
  Profiles with a comprehensive set of genetic variants to look for markers implicated in response to Mastiha treatment.
Metabolomic profile | 6 months
  Quantification of endogenous metabolites from different compound classes
Metagenomic profile | 6 months
  Association of gut microbes with Mastiha treatment in NAFLD
Epigenetic profile | 6 months
  Identification of the subset of variably methylated regions with low within-individual variability over the six months period of the study to correlate them to treatment.
Effect of Mastiha on different BMI categories | 6 months
  Identification of the effect of Mastiha on different obesity categories: Class I obesity (BMI ≤ 35) and Class II or III obesity (BMI> 35)

CONTACTS AND LOCATIONS:
Overall Officials: G V DEDOUSIS, PROF., Study Director — Harokopio University
Locations (1):
- Harokopio University, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pavlides M, Banerjee R, Sellwood J, Kelly CJ, Robson MD, Booth JC, Collier J, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging predicts clinical outcomes in patients with chronic liver disease. J Hepatol. 2016 Feb;64(2):308-315. doi: 10.1016/j.jhep.2015.10.009. Epub 2015 Nov 10. PMID 26471505
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Hassan K, Bhalla V, El Regal ME, A-Kader HH. Nonalcoholic fatty liver disease: a comprehensive review of a growing epidemic. World J Gastroenterol. 2014 Sep 14;20(34):12082-101. doi: 10.3748/wjg.v20.i34.12082. PMID 25232245
- [Background] Abenavoli L, Milic N, Di Renzo L, Preveden T, Medic-Stojanoska M, De Lorenzo A. Metabolic aspects of adult patients with nonalcoholic fatty liver disease. World J Gastroenterol. 2016 Aug 21;22(31):7006-16. doi: 10.3748/wjg.v22.i31.7006. PMID 27610012
- [Background] Yao H, Qiao YJ, Zhao YL, Tao XF, Xu LN, Yin LH, Qi Y, Peng JY. Herbal medicines and nonalcoholic fatty liver disease. World J Gastroenterol. 2016 Aug 14;22(30):6890-905. doi: 10.3748/wjg.v22.i30.6890. PMID 27570425
- [Background] Dongiovanni P, Romeo S, Valenti L. Genetic Factors in the Pathogenesis of Nonalcoholic Fatty Liver and Steatohepatitis. Biomed Res Int. 2015;2015:460190. doi: 10.1155/2015/460190. Epub 2015 Jul 27. PMID 26273621
- [Background] Fan JG, Cao HX. Role of diet and nutritional management in non-alcoholic fatty liver disease. J Gastroenterol Hepatol. 2013 Dec;28 Suppl 4:81-7. doi: 10.1111/jgh.12244. PMID 24251710
- [Background] Triantafyllou A, Chaviaras N, Sergentanis TN, Protopapa E, Tsaknis J. Chios mastic gum modulates serum biochemical parameters in a human population. J Ethnopharmacol. 2007 Apr 20;111(1):43-9. doi: 10.1016/j.jep.2006.10.031. Epub 2006 Nov 6. PMID 17150319
- [Derived] Kanoni S, Kumar S, Amerikanou C, Kurth MJ, Stathopoulou MG, Bourgeois S, Masson C, Kannt A, Cesarini L, Kontoe MS, Milanovic M, Roig FJ, Beribaka M, Campolo J, Jimenez-Hernandez N, Milosevic N, Llorens C, Smyrnioudis I, Francino MP, Milic N, Kaliora AC, Trivella MG, Ruddock MW, Medic-Stojanoska M, Gastaldelli A, Lamont J, Deloukas P, Dedoussis GV, Visvikis-Siest S. Nutrigenetic Interactions Might Modulate the Antioxidant and Anti-Inflammatory Status in Mastiha-Supplemented Patients With NAFLD. Front Immunol. 2021 May 7;12:683028. doi: 10.3389/fimmu.2021.683028. eCollection 2021. PMID 34025683